CLINICAL TRIAL: NCT02110186
Title: A Prospective, Comparative Study to Evaluate Effectiveness and Safety of Dynamic Stabilization in Treatment of Lumbar Disc Herniation
Brief Title: Lumbar Intervertebral Disc Herniation
Acronym: LIDH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Qiang Zhou, MD. PhD., Deputy Chair of the Department of Orthopedics, Chair of the Department of Spine Surgical Group, Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMMU-ORTHO-2012-001
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Lumbar Disc Herniation
Keywords: lumbar disc herniation; dynamic stabilization; discectomy with posterior dynamic stabilization; discectomy alone; discectomy with internal fixation and fusion
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Diskectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Discectomy and dynamic stabilization (Experimental): Discectomy with posterior dynamic stabilization
  Interventions: Device: Dynamic Stabilization; Procedure: Discectomy
- Discectomy alone (Active Comparator): Discectomy
  Interventions: Procedure: Discectomy
- Discectomy and fusion (Active Comparator): Discectomy with internal fixation and fusion
  Interventions: Procedure: Discectomy; Device: Instrumentation and fusion

INTERVENTIONS:
Device: Dynamic Stabilization
  Arms: Discectomy and dynamic stabilization
Procedure: Discectomy
Device: Instrumentation and fusion
  Arms: Discectomy and fusion

SUMMARY:
The purpose of this study is to compare safety and outcomes of the following treatments of lumbar disc herniation: (1) discectomy with posterior dynamic stabilization with those of (2) discectomy alone or (3) discectomy with internal fixation and fusion.

Discectomy with posterior dynamic stabilization is proposed as the most effective treatment to improve range of motion, and to be similarly effective to discectomy alone and discectomy with internal fixation and fusion for other functional outcomes after surgery.

DETAILED DESCRIPTION:
The purpose of this study is to compare outcomes of (1) discectomy with posterior dynamic stabilization with those of (2) discectomy alone or (3) discectomy with internal fixation and fusion.

Study aims are:

1. To demonstrate superiority of discectomy with posterior dynamic stabilization over discectomy alone and discectomy with internal fixation and fusion in range of motion at the operated level;
2. To demonstrate non-inferiority of discectomy with posterior dynamic stabilization compared to discectomy alone and discectomy with internal fixation and fusion in functional outcomes as measured by change in Oswestry Disability Index;
3. To compare radiological, clinical, patient-reported and safety outcomes among the three surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age between 20 and 60 years inclusive
* Radiographic evidence of single level lumbar disc herniation
* Scheduled for single-level lumbar discectomy with or without fusion or dynamic stabilization
* Preoperative ODI ≥ 30
* Clinical symptoms consistent with lumbar disc herniation determined by history or physical exam:

  * Radicular back or lower extremity pain and/or
  * Decreased muscular strength and/or
  * Abnormal sensation
* Involved disk at the spinal level between L2 and S1
* Failed to gain adequate symptom relief from at least one month of adequate non-operative treatment, except in patients with severe symptoms that require immediate surgery (at surgeon's discretion)
* Absence of significant symptomatic adjacent segment disk herniation

Exclusion Criteria:

* Cauda equine syndrome
* Previous spinal surgery, except previous discectomy at the same segment
* Patients with other lumbar conditions that will, in the opinion of the investigator, interfere with clinical outcomes (e.g. spinal structural deformities, spinal fractures, ankylosing spondylitis, spinal tuberculosis, spinal infection, spinal tumors, symptomatic cervical spinal disease)
* Osteoporosis defined as T-score ≤ -2.5. BMD will be measured by DEXA performed on lumbar spine
* Systemic infection such as AIDS, HIV, and active hepatitis
* Recent history (less than 3 years) of chemical substance dependency or significant psychosocial disturbance, which may impact the outcome or study participation
* Participation in a clinical trial of another investigational drug or device within the past 30 days

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 195 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-07 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Range of motion in sagittal plane at the operated level | 24 months
Mean Change in Oswestry Disability Index (ODI) | Baseline, 24 months

SECONDARY OUTCOMES:
Change in Lumbar Pain Numeric Rating Scale (NRS) | Baseline, 24 months
Change in Leg Pain NRS | Baseline, 24 months

OTHER OUTCOMES:
Change in SF-36 dimensions | Baseline, 24 Months
Radiographic Evaluations | 24 months
Time to occurrence and relationship to surgery of adverse events | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Military Medical University/Southwest Hospital, Chongqing, China